CLINICAL TRIAL: NCT00440089
Title: Effects of Hands-on-Healing vs. Touch for Fatigue and Inflammation in Breast Cancer Survivors
Brief Title: Effects of Hands-on-Healing vs. Touch for Fatigued Breast Cancer Survivors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Shamini Jain, University of California San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: F31AT003021 (NIH); F31AT003021 (NIH)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: Cancer; Fatigue; Breast Cancer; Healing; Energy Healing; Complementary; Alternative; Immune; Cytokine; Hormone; Cortisol; Placebo; Mock Healing
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: Hands-on-Healing

SUMMARY:
This randomized controlled trial examines the efficacy of hands-on-healing for fatigue and immune function in breast cancer survivors. Participants may be randomized to one of three groups: hands-on-healing, touch alone, or a control group.

DETAILED DESCRIPTION:
Please see our website at http://healing.ucsd.edu for detailed information on the study.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal and postmenopausal women between the ages of 18 to 70 years.
* Ability to give informed consent.
* Breast cancer survivors who have undergone surgery, including lumpectomy and simple or total mastectomy, followed by chemotherapy or a combination of chemo- and radio-therapy. We have elected to study survivors instead of patients actively undergoing treatment to alleviate subject burden and risk during this protocol.
* Stage I to III breast cancer survivors.
* Breast cancer survivors who have finished their chemotherapy and/or radiotherapy at least one month prior to 60 months prior.
* Breast cancer survivors with above-normative levels of fatigue.

Exclusion Criteria:

* Breast cancer patients who are currently receiving or who are scheduled to receive radiation or chemotherapy during the course of this intervention study.
* Patients with current major depression, current or history of prior bipolar illness, currently on psychotropic medications.
* Patients with other diseases that are known to induce fatigue (e.g., thyroid disorder; sleep disorders).
* Patients with other inflammatory diseases that affect cytokine levels.
* Patients with a history of other cancers, and stage IV breast cancer.
* Patients undergoing current chemotherapy and/or radiotherapy.
* Men with breast cancer.
* Substance abuse/dependence.
* Continued use of another biofield-based intervention (e.g., Reiki, Qi-Gong, Healing Touch, Therapeutic Touch, Johrei).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Multiple Fatigue Symptom Inventory

SECONDARY OUTCOMES:
Inflammatory Immune Markers
Diurnal Cortisol Variability

CONTACTS AND LOCATIONS:
Overall Officials: Shamini Jain, Ph.D., Principal Investigator — University of California, Los Angeles; Paul J Mills, Ph.D., Principal Investigator — UCSD School of Medicine
Locations (2):
- United States (2):
  - Clinical Research Center, UCSD Campus, La Jolla, California
  - General Clinical Research Center, UCSD Medical Center, San Diego/Hillcrest, California